CLINICAL TRIAL: NCT07269860
Title: The Impact of Osteopathic Manipulative Medicine on Radiotracer and Isosulfan Blue Dye Uptake During Breast Conserving Surgery and Sentinel Lymph Node Biopsy.
Brief Title: Impact of Osteopathic Manipulative Medicine on Sentinal Lymph Node Biopsy Dye and Tracer Uptake
Acronym: OMM on SLNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Tucson Osteopathic Medical Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00004477
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Osteopathic Manipulative Medicine; Sentinal lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to receive standard of care or intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage (No Intervention): Patients will receive the standard of care practice for SLNB of 9 minutes of circular massage over the nipple areolar complex to disperse isosulfan blue dye and radiotracer that were injected into the breast.
- OMM + Massage (Experimental): 5 min of massage plus perform osteopathic techniques including 1 minute of each of the following: opening the thoracic inlet, pectoral traction, and axillary pump. Thoracic pump will be done for 2 minutes. Isosulfan blue dye and radiotracer will then be injected followed by massage as done in the current standard of practice. The injection and massage are performed as per standard of care.
  Interventions: Procedure: OMM prior to SLNB

INTERVENTIONS:
Procedure: OMM prior to SLNB — Perform osteopathic techniques including 1 minute of each of the following: opening the thoracic inlet, pectoral traction, and axillary pump. Thoracic pump will be done for 2 minutes. Isosulfan blue dye and radiotracer will then be injected followed by massage as done in the current standard of practice. The injection and massage are performed as per standard of care.
  Arms: OMM + Massage

SUMMARY:
The goal of this clinical trial is to learn if osteopathic manipulative medicine (OMM) will allow for more uptake of isosulfan blue dye and radiotracers used in sentinal lymph node biopsy (SLNB) compared to massage alone. SLNB is used to characterize the stage and spread of cancer cells in breast cancer patients. The main questions it aims to answer is:

- Does OMM + massage allow for greater uptake of isosulfan blue dye and radiotracer in the lymph nodes compared to current standard of practice of breast massage after isosulfan blue dye and radiotracer injection.

Researchers will compare OMM + massage to current standard of practice of breast massage.

Randomization: Patients will be randomized prior to surgical intervention as to which arm of the study they will be assigned to: Massage (current standard) vs OMM + Massage

Massage: 9 minutes of circular massage over the nipple areolar complex to disperse isosulfan blue dye and radiotracer that were injected into the breast. Massage following injection is standard of care.

OMM+ Massage: 5 minutes of massage as above and then will perform osteopathic techniques including 1 minute of each of the following: opening the thoracic inlet, pectoral traction, and axillary pump. Thoracic pump will be done for 2 minutes. Isosulfan blue dye and radiotracer will then be injected followed by massage as done in the current standard of practice. The injection and massage are performed as per standard of care.

DETAILED DESCRIPTION:
In order to appropriately and adequately treat breast cancer, sentinel lymph node mapping and biopsies are used to characterize stage and spread of cancer cells. Isosulfan blue dye and radiotracers are used to identify and target the sentinel lymph node and, therefore the specific group of lymphatic vessels that are draining the breast cancer. In order to identify the sentinel node, lymphatic vessels must be draining properly to allow for dye or radiotracer to have adequate uptake within the lymphatic system. Lymphatic vessels themselves or the fascia surrounding lymphatic vessels can have innate or pathological dysfunction that can be improved by osteopathic manipulation of these structures allowing for more accurate node identification with blue dye and radiotracer.

This study will look at the impact of osteopathic manipulation on fascia of the anterior chest wall as well as the lymphatic system draining the breast. We will compare the current standard of practice of breast massage after isosulfan blue dye and radiotracer injection to OMM + massage. Qualitative blue dye uptake in the sentinel lymph node as well as target values of radiotracer will be analyzed.

Two main points of data will be collected in order to determine how well the axilla mapped for that operation. These data points are the amount of isosulfan blue dye uptake in the lymph nodes and the target values on the neoprobe that tell how much radio tracer made it to those lymph nodes. The more blue in color a lymph node is and the higher the target value on the neoprobe determines if a node is the sentinel node in a typical breast cancer operation. We will use those same end points to assess if we have better uptake of blue dye or radio tracer in the axilla with or without the addition of OMM. In order to quantify the amount of blue dye uptake in a node, each node removed during the procedure will be categorized under blue or not blue. For those nodes that are blue, they will be analyzed as falling under 100%, 75%, 50%, or 25% blue. Meaning if half of the node is blue and half is a normal tissue color, this node would count under the 50% blue category. All blue nodes are typically removed during a sentinel lymph node operation. The second endpoint is the target value. The neoprobe detects and quantifies the amount of the radiotracer that was previously injected. If a node uptakes the radiotracer, it will be detected with the neoprobe. In a typical sentinel node operation, the nodes with the most tracer signal are removed and the target value (10 second count of the amount of radiotracer) is obtained for that node. Any other node in the axilla that is 10% of that highest target value will also be removed as it has the chance of being the sentinel node. For example if the hottest node in the axilla has a target value of 15000 then any node that is detected to have a value of 1500 or higher via the neoprobe will be removed. All radioactive nodes that fall into this 10% rule will be removed as per the usual surgery protocol and a target value obtained for each node. These values will be recorded as a way to determine how effective the radiotracer uptake was in the axilla.

Hypothesis: OMM + massage will have increased radiotracer target values and more isosulfan blue dye uptake in the sentinel lymph node compared to massage alone.

ELIGIBILITY:
Inclusion Criteria:

* First time breast cancer patients (female only) undergoing breast conserving surgery (lumpectomy or partial mastectomy) and sentinel lymph node biopsy.

Exclusion Criteria:

* Previous breast cancer
* previous axillary surgery
* previous chest wall or axillary radiation
* previous breast surgery
* known axillary disease
* patients undergoing total mastectomies

Contraindications to OMM include inability to access the axilla due to range of motion, previous shoulder injury or shoulder surgery on the treatment side, fractures or metastatic lesions to the bones on the treatment side, open wounds over the treatment area or underlying abscess/infection, pacemaker on the side of treatment, subclavian vein central line or port.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — First time breast cancer patients (female only) undergoing breast conserving surgery (lumpectomy or partial mastectomy) and sentinel lymph node biopsy.
Enrollment: 27 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of isosulfan blue dye uptake in the lymph nodes | Through study completion, 4 months
  In order to quantify the amount of blue dye uptake in a node, each node removed during the procedure will be categorized under blue or not blue. The percentage of blue dye uptake is determined visually by the operating surgeon. All surgeons were trained on how to identify these percentages. A node is labeled as 25% blue if it had a blue channel and/or minimal blue coloration of the node, 50% blue if it is a moderately/partially blue node, 75% blue if it was a mostly blue node, and 100% blue if it was a completely blue node.

SECONDARY OUTCOMES:
Target value of neoprobe that tell how much radiotracer makes it to the lymph nodes | Through study completion, 4 months
  The second endpoint is the target value. The neoprobe detects and quantifies the amount of the radiotracer that was previously injected. If a node uptakes the radiotracer, it will be detected with the neoprobe. In a typical sentinel node operation, the nodes with the most tracer signal are removed and the target value (10 second count of the amount of radiotracer) is obtained for that node. Any other node in the axilla that is 10% of that highest target value will also be removed as it has the chance of being the sentinel node. For example if the hottest node in the axilla has a target value of 15000 then any node that is detected to have a value of 1500 or higher via the neoprobe will be removed. All radioactive nodes that fall into this 10% rule will be removed as per the usual surgery protocol and a target value obtained for each node. These values will be recorded as a way to determine how effective the radiotracer uptake was in the axilla.

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Stejskal, DO, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center - Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No